CLINICAL TRIAL: NCT07021729
Title: Comparison of Conventional Clarithromycin Vs Alternative Levofloxacin Based Regimen in Treatment of Helicobacter Pylori Infection
Brief Title: Comparison of Two Treatment Regimens of Helicobacter Pylori Infection
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rehman Medical Institute - RMI (Other)
Responsible Party: Principal Investigator, Wajeeha Qayyum, Consultant/Assistant Professor Medicine, Rehman Medical Institute - RMI
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMI/RMI-REC/approval/181
Record Dates: First submitted 2023-08-17; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Helicobacter Pylori Infection
Keywords: clarithromycin; levofloxacin; helicobacter pylori
MeSH Terms: interventions — Clarithromycin; Metronidazole; Omeprazole; Levofloxacin; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regime 1 (Active Comparator): This arm will receive clarithromycin based regimen for eradication of H pylori infection (as per approved guidelines)
  Interventions: Drug: Clarithromycin
- Regime 2 (Active Comparator): This arm will receive levofloxacin based regimen for eradication of H pylori infection (as per approved guidelines)
  Interventions: Drug: Levofloxacin

INTERVENTIONS:
Drug: Clarithromycin — Drug regimens will be given for 14 days, and omeprazole for 6weeks
  Other Names: Metronidazole; omeprazole
  Arms: Regime 1
Drug: Levofloxacin — Drug regimens will be given for 14 days, and omeprazole for 6weeks
  Other Names: amoxicillin; omeprazole
  Arms: Regime 2

SUMMARY:
The goal of this interventional study is to compare the efficacy of clarithromycin Vs levofloxacin based regimen in treatment of Helicobacter pylori infection in patients presenting to medical OPD who are tested positive for H pylori infection.. The main question[s] it aims to answer are:

• Which regimen is superior in terms of efficacy Participants will be treated for H pylori Infection in with two different regimen If there is a comparison group: Researchers will compare two groups Group 1 will receive clarithromycin based regimen group 2 will receive levofloxacin based regimen to see the treatment response.

DETAILED DESCRIPTION:
This interventional study will be conducted in department of medicine, Rehman Medical Institute, Peshawar.

Study duration: 10 months after the issuance of ethical approval Sample size: Sample size is calculated using a two-tailed alpha test with a significance level of 0.05 and 90% power to detect 23% difference in the eradication rate of the two regimens. The total number of patients required to prove the hypothesis is 156, 78 in each group.

Study population: Patients coming to OPD with symptoms suggestive of H pylori infection will undergo screening by Hpylori stool antigen. If it comes to be positive then they will be enrolled in study after applying inclusion/exclusion criteria.

Inclusion criteria: All patients who tested positive on stool antigen will be included. Age >12 years and both genders will be included.

Exclusion criteria: patients under 12 years old. Patients who have penicillin allergy.

Patients who have underlying dysrhythmia forbidding the use of macrolide. Patient who have hypersensitivity to any of these antibiotics.

Study population will be divided in two groups. Group 1 will receive regimen number 1 and group 2 will receive regimen number 2.( regimens are described below.) Regimen 1 (R1): Clarithromycin 500mg BD, plus metronidazole 400mg TDS for 14days and Omeprazole 40mg BD for 6 weeks.

Regimen 2(R2): Levofloxacin 500mg OD plus Amoxicillin 1gm BD for 14 days and omeprazole 40mg Bd for 6 weeks.

The patients will be followed 2 weeks after completion of treatment. On follow up, their symptoms improvement, compliance and side effects will be documented. They will undergo stool Ag test again to assess treatment response.

ELIGIBILITY:
Inclusion Criteria:

* All patients who tested positive on stool antigen will be included.

Exclusion Criteria:

* patients under 12 years old. Patients who have penicillin allergy.
* Patients who have underlying dysrhythmia forbidding the use of macrolide.
* Patient who have hypersensitivity to any of these antibiotics.

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Treatment of H pylori infection | 2weeks after completion of treatment regimen
  Treatment of H pylori infection documented by negative stool antigen

CONTACTS AND LOCATIONS:
Overall Officials: Wajeeha Qayyum, FCPS, Principal Investigator — Rehman Medical Institute

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Hooi JKY, Lai WY, Ng WK, Suen MMY, Underwood FE, Tanyingoh D, Malfertheiner P, Graham DY, Wong VWS, Wu JCY, Chan FKL, Sung JJY, Kaplan GG, Ng SC. Global Prevalence of Helicobacter pylori Infection: Systematic Review and Meta-Analysis. Gastroenterology. 2017 Aug;153(2):420-429. doi: 10.1053/j.gastro.2017.04.022. Epub 2017 Apr 27. PMID 28456631
- [Background] Sugano K, Tack J, Kuipers EJ, Graham DY, El-Omar EM, Miura S, Haruma K, Asaka M, Uemura N, Malfertheiner P; faculty members of Kyoto Global Consensus Conference. Kyoto global consensus report on Helicobacter pylori gastritis. Gut. 2015 Sep;64(9):1353-67. doi: 10.1136/gutjnl-2015-309252. Epub 2015 Jul 17. PMID 26187502
- [Background] 4. Shah SRH, , Almugadam BS, Hussain Akbar, Ahmad T, Ahmed S , Sadiqui S. Epidemiology and risk factors of Helicobacter pylori infection in Timergara city of Pakistan: A cross-sectional study. Clinical Epidemiology and Global Health 12 (2021) 100909.
- [Background] Azab ET, Thabit AK, McKee S, Al-Qiraiqiri A. Levofloxacin versus clarithromycin for Helicobacter pylori eradication: are 14 day regimens better than 10 day regimens? Gut Pathog. 2022 Jun 6;14(1):24. doi: 10.1186/s13099-022-00502-3. PMID 35668511
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Gisbert JP, Kuipers EJ, Axon AT, Bazzoli F, Gasbarrini A, Atherton J, Graham DY, Hunt R, Moayyedi P, Rokkas T, Rugge M, Selgrad M, Suerbaum S, Sugano K, El-Omar EM; European Helicobacter and Microbiota Study Group and Consensus panel. Management of Helicobacter pylori infection-the Maastricht V/Florence Consensus Report. Gut. 2017 Jan;66(1):6-30. doi: 10.1136/gutjnl-2016-312288. Epub 2016 Oct 5. PMID 27707777
- [Background] Rizwan M, Fatima N, Alvi A. Epidemiology and pattern of antibiotic resistance in Helicobacter pylori: scenario from Saudi Arabia. Saudi J Gastroenterol. 2014 Jul-Aug;20(4):212-8. doi: 10.4103/1319-3767.136935. PMID 25038206
- [Background] Haji-Aghamohammadi AA, Bastani A, Miroliaee A, Oveisi S, Safarnezhad S. Comparison of levofloxacin versus clarithromycin efficacy in the eradication of Helicobacter pylori infection. Caspian J Intern Med. 2016 Fall;7(4):267-271. PMID 27999644
- [Background] Sebghatollahi V, Soheilipour M, Khodadoostan M, Shavakhi A, Shavakhi A. Levofloxacin-containing versus Clarithromycin-containing Therapy for Helicobacter pylori Eradication: A Prospective Randomized Controlled Clinical Trial. Adv Biomed Res. 2018 Mar 27;7:55. doi: 10.4103/abr.abr_133_17. eCollection 2018. PMID 29657940